CLINICAL TRIAL: NCT05965076
Title: Analysis of the Effectiveness of the Use of Glycine Powder and Angled Implant Brush in Oral Hygiene Maintenance in Patients Reinstated With Columbus Bridge ProtocolTM: a Factorial Randomized Study
Brief Title: Analysis of the Effectiveness of the Use of Glycine Powder and Angled Implant Brush in Oral Hygiene Maintenance in Patients Reinstated With Columbus Bridge ProtocolTM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Crupi Armando, Principal investigator, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 99110619
Record Dates: First submitted 2023-07-06; First posted 2023-07-28 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Plaque, Dental
Keywords: glycine; airflow; full-arch; angled toothbrush
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard (Active Comparator): Patients will be professionally treated with standard dental hygiene treatment, and they will use a standard toothbrush for their domiciliary oral hygiene.
  Interventions: Procedure: Standard Professional Oral Hygiene; Behavioral: Standard Domiciliary Oral Hygiene
- Glycine (Experimental): Patients will be professionally treated by adding glycine perio-flow in the treatment, and they will use a standard toothbrush for their domiciliary oral hygiene.
  Interventions: Procedure: Glycine Perio Flow; Behavioral: Standard Domiciliary Oral Hygiene
- Angled toothbrush (Experimental): Patients will be professionally treated with standard dental hygiene treatment, and they will use an angled toothbrush for their domiciliary oral hygiene.
  Interventions: Behavioral: Angled Toothbrush; Procedure: Standard Professional Oral Hygiene
- Glycine - Angled toothbrush (Experimental): Patients will be professionally treated by adding glycine perio-flow in the treatment, and they will use an angled toothbrush for their domiciliary oral hygiene.
  Interventions: Procedure: Glycine Perio Flow; Behavioral: Angled Toothbrush

INTERVENTIONS:
Procedure: Glycine Perio Flow — Professional plaque and tartar removal by means of titanium curettes, bridge and implant floss and glycine perio-flow.
  Arms: Glycine; Glycine - Angled toothbrush
Behavioral: Angled Toothbrush — Patients will be educated and motivated in domiciliary oral hygien by means of bridge and implant floss and an angled toothbrush.
  Arms: Angled toothbrush; Glycine - Angled toothbrush
Procedure: Standard Professional Oral Hygiene — Professional plaque and tartar removal by means of titanium curettes, bridge and implant floss.
  Arms: Angled toothbrush; Standard
Behavioral: Standard Domiciliary Oral Hygiene — Patients will be educated and motivated in domiciliary oral hygien by means of bridge and implant floss and a standard toothbrush.
  Arms: Glycine; Standard

SUMMARY:
This study aims at comparing different procedures of Professional Oral Hygiene (POH) and Domiciliary Oral Hygiene (DOH) in Columbus Bridge ProtocolTM full-arch reinstated patients by dividing a sample of at least 74 patients into 4 groups with a 1:1:1:1 ratio. The patients will randomly be assigned to a "Standard" or "Glycine Perio Flow" Professional treatment, and to a "Standard" or "Angled" Toothbrush for their Domiciliary oral hygiene.

Data about bacterial plaque presence is collected both before and after unscrewing the denture, when it comes to implant abutments. Instead, Denture Plaque Index will be collected after unscrewing the denture, by means of erythrosine and analyzed using a specific software that allows to compute the percentage of plaque on the denture.

Patients will be seen after 3 months in order to figure out differences between DOH groups, by measuring plaque on abutments and on the denture after unscrewing it.

At the moment there are no scientific studies trying to determine which professional and domiciliary procedures might be more efficient to control bacterial plaque in Columbus Bridge ProtocolTM reinstated patients.

Statistically significant lower Plaque Index (PI) and Denture Plaque Index (DPI) scores are expected in patients treated with glycine perio flow, compared to standard treated patients. However, when it comes to angled toothbrush, lower PI and DPI are expected not to be statistically significant.

Expectation from this study is to get information on how to improve full-arch patients' therapy in order to reduce peri-implant diseases which are related to bacterial plaque.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18years
* Good systemic health, with ASA classification <= 2
* Columbus Bridge ProtocolTM reinstation from at least six months

Exclusion Criteria:

* Heavy smokers (>= 10 cigarettes per day)
* Pregnancy or breastfeeding
* Autoimmune diseases with or without oral involvement
* Biological complications on at least one of the dental implants
* Perimplantits diagnosis, defined according to Lindhe et al's criteria [5]
* Radicular bone <4mm, evaluated by means of RX
* Use of gingival overgrowth inducing drugs
* Cognitive or motor impairments
* Full-arch reinstations performed in other structures
* Respiratory issues
* Infective diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Denture Plaque Index (DPI) | T0: first session (for professional oral hygiene).
  This study's primary outcome is the plaque index on the denture (DPI). Plaque indexes will be determined by means of erythrosine (GC Tri Plaque ID GelTM, Tokyo, Japan).
  Pictures in jpg format will be taken with a digital Nikon D80 camera with 105mm macro lens and processed with ImageJ 1.45s software (National Institutes of Health, Bethesda, MD, USA). Pictures will be converted into binary monochrome images. Specific standard thresholds will be determined to differentiate the plaque pixels (blue) from the plaque free ones (pink). This procedure is already proven by literature.
Denture Plaque Index (DPI) | T1: second session, after 3 months (for domiciliary oral hygiene).
  This study's primary outcome is the plaque index on the denture (DPI). Plaque indexes will be determined by means of erythrosine (GC Tri Plaque ID GelTM, Tokyo, Japan).
  Pictures in jpg format will be taken with a digital Nikon D80 camera with 105mm macro lens and processed with ImageJ 1.45s software (National Institutes of Health, Bethesda, MD, USA). Pictures will be converted into binary monochrome images. Specific standard thresholds will be determined to differentiate the plaque pixels (blue) from the plaque free ones (pink). This procedure is already proven by literature.

SECONDARY OUTCOMES:
Probing Depth (PD); | T0: first session (for professional oral hygiene).
  Periodontal indexes will be determined on four areas for each implant by means of a UNC 15 (Hu-Friedy, Chicago, IL, USA) Probe. Probing depth is evaluated in mm.
Probing Depth (PD); | T1: second session, after 3 months (for domiciliary oral hygiene).
  Periodontal indexes will be determined on four areas for each implant by means of a UNC 15 (Hu-Friedy, Chicago, IL, USA) Probe. Probing depth is evaluated in mm.
Bleeding on Probing (BoP); | T0: first session (for professional oral hygiene).
  Periodontal indexes will be determined on four areas for each implant by means of a UNC 15 (Hu-Friedy, Chicago, IL, USA) Probe. Bleeding on probing is evaluated as presence of bleeding (yes/no).
Bleeding on Probing (BoP); | T1: second session, after 3 months (for domiciliary oral hygiene).
  Periodontal indexes will be determined on four areas for each implant by means of a UNC 15 (Hu-Friedy, Chicago, IL, USA) Probe. Bleeding on probing is evaluated as presence of bleeding (yes/no).
Plaque Index on implant abutments | T0: first session (for professional oral hygiene).
  Periodontal indexes will be determined on four areas for each implant by means of a UNC 15 (Hu-Friedy, Chicago, IL, USA) Probe. PI is defined as plaque presence (yes/no) on the abutment or denture by means of erythrosine gel.
Plaque Index on implant abutments | T1: second session, after 3 months (for domiciliary oral hygiene).
  Periodontal indexes will be determined on four areas for each implant by means of a UNC 15 (Hu-Friedy, Chicago, IL, USA) Probe. PI is defined as plaque presence (yes/no) on the abutment or denture by means of erythrosine gel.

CONTACTS AND LOCATIONS:
Locations (1):
- S.C. Riabilitazione Orale Protesi Maxillo-Facciale e Implantologia Dentaria, Torino, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Lindhe J, Meyle J; Group D of European Workshop on Periodontology. Peri-implant diseases: Consensus Report of the Sixth European Workshop on Periodontology. J Clin Periodontol. 2008 Sep;35(8 Suppl):282-5. doi: 10.1111/j.1600-051X.2008.01283.x. PMID 18724855
- [Result] Abi Nader S, Eimar H, Momani M, Shang K, Daniel NG, Tamimi F. Plaque Accumulation Beneath Maxillary All-on-4 Implant-Supported Prostheses. Clin Implant Dent Relat Res. 2015 Oct;17(5):932-7. doi: 10.1111/cid.12199. Epub 2014 Jan 27. PMID 24461161
- [Result] Mensi M, Scotti E, Sordillo A, Agosti R, Calza S. Plaque disclosing agent as a guide for professional biofilm removal: A randomized controlled clinical trial. Int J Dent Hyg. 2020 Aug;18(3):285-294. doi: 10.1111/idh.12442. Epub 2020 May 26. PMID 32348624